CLINICAL TRIAL: NCT04481724
Title: Effects of Gamma-linolenic Acid Supplementation on Weight Loss Maintenance in the Virta Treatment
Brief Title: Gamma-linolenic Acid Supplementation Study
Acronym: GLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virta Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-6
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Weight Trajectory
MeSH Terms: conditions — Body-Weight Trajectory | interventions — gamma-Linolenic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 3:1, GLA:placebo. Interim analyses of the primary outcome will be performed at 12 and 18 months; if greater weight loss is maintained in the GLA compared to placebo group, the study will be unblinded and placebo group participants will cross over to the GLA group for the remainder of the trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gamma-linolenic acid (GLA) supplementation (Experimental): Sonova GLA safflower oil (840 mg GLA per day)
  Interventions: Dietary Supplement: gamma-linolenic acid
- placebo control (Placebo Comparator): 1500 mg 'light' olive oil per day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: gamma-linolenic acid — 3 capsules per day of GLA for 24 months
  Arms: gamma-linolenic acid (GLA) supplementation
Dietary Supplement: placebo — 3 capsules per day of placebo for 24 months
  Arms: placebo control

SUMMARY:
Weight regain following weight loss is common. In rodent models of obesity and pilot studies in humans, increasing membrane arachidonic acid content improves fuel partitioning and prevents weight regain. This study aims to understand the effect of gamma-linolenic acid (GLA) supplementation on weight loss maintenance in Virta Health patients.

DETAILED DESCRIPTION:
The primary purpose of this research is to determine if GLA supplementation reduces weight regain over 24 months in Virta Health patients.

The secondary purpose is to determine the effect of GLA supplementation on diabetes-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 yrs
* Patients referred to Virta Health by employers or insurers
* Weight loss greater than or equal to 7% of initial weight and current BMI > 25 kg/m2
* Willing to take 3 supplement capsules daily
* Able to understand study procedures and willing to provide informed consent
* English-speaking

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients who are taking or are prescribed orlistat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Difference in change in body weight between groups over time | 0, 12, 18, and 24 months
  Body weight measured on a calibrated scale. Interim analyses at 12 and 18 months; if greater weight loss is maintained in the GLA compared to placebo group, the study will be unblinded and placebo group participants will cross over to GLA for the remainder of the trial.

SECONDARY OUTCOMES:
Difference in subjective neuropathy symptoms between groups over time | 0, 6, 12, 18, and 24 months
  Michigan Neuropathy Screening Instrument (MNSI) administered every 6 months
Difference in health-related quality of life between groups over time | 0, 6, 12, 18, and 24 months
  Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) administered every 6 months
Difference in perceived control over eating between groups over time | 0, 6, 12, 18, and 24 months
  Eating Loss of Control Scale (ELOCS) administered every 6 months
Difference in body image and satisfaction between groups over time | 0, 6, 12, 18, and 24 months
  Body Image States Scale (BISS) administered every 6 months
Difference in medication prescriptions between groups over time | 0, 6, 12, 18, and 24 months
  Prescribed medications obtained from medical record
Difference in hemoglobin A1c between groups over time | Approximately 0, 6, 12, 18, and 24 months
Difference in ketones between groups over time | 0, 6, 12, 18, and 24 months
  Finger prick ketone values
Difference in blood glucose between groups over time | 0, 6, 12, 18, and 24 months
  Finger prick glucose values

CONTACTS AND LOCATIONS:
Overall Officials: Shaminie Athinarayanan, PhD, Principal Investigator — Virta Health; Rebecca Adams, PhD, Study Director — Virta Health
Locations (1):
- Virta Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiers will be removed and data could then be used for future research studies or distributed to another investigator for future research studies without additional informed consent.